CLINICAL TRIAL: NCT06674460
Title: Treatment of Acute Ischemic Stroke With Edaravone Dexborneol Sublingual Tablets in Small Vessel Disease: A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Treatment of Acute Ischemic Stroke With Edaravone Dexborneol Sublingual Tablets in Small Vessel Disease
Acronym: TASTE-SVD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASTE-SVD; 2023ZD0504900 (Other Grant/Funding Number: National Science and Technology Major Project)
Record Dates: First submitted 2024-10-23; First posted 2024-11-05 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Cerebral Small Vessel Disease; Ischemic Stroke
Keywords: sublingual edaravone dexborneol; cerebral small vessel disease; acute ischemic cerebral small vessel disease; cognition
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone Dexborneol Sublingual Tablets (Experimental): One tablet of Edaravone Dexborneol Sublingual Tablet (containing 30mg Edaravone and 6mg Dexborneol) to be taken sublingually, twice daily.
  Interventions: Drug: Edaravone Dexborneol Sublingual Tablets
- Placebo (Placebo Comparator): One placebo tablet, to be taken sublingually, twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edaravone Dexborneol Sublingual Tablets — One tablet of Edaravone Dexborneol Sublingual Tablet (containing 30mg Edaravone and 6mg Dexborneol) to be taken sublingually, twice daily.
  Arms: Edaravone Dexborneol Sublingual Tablets
Drug: Placebo — One placebo tablet, to be taken sublingually, twice daily
  Arms: Placebo

SUMMARY:
This study is a multicenter, randomized, double-blind, placebo-controlled trial designed to evaluate the efficacy and safety of Edaravone Dexborneol Sublingual Tablets in patients with acute ischemic stroke due to small vessel disease (TASTE-SVD).

The study will enroll approximately 600 participants aged 30 to 80 years who have experienced a recent small subcortical infarct (RSSI) confirmed by MRI. Participants will be randomized in a 1:1 ratio into either the Edaravone Dexborneol Sublingual Tablets group or the placebo group, with a 24-week treatment period followed by a 28-week follow-up.

The primary endpoint is a hierarchical composite endpoint at week 24, including all-cause mortality, modified Rankin Scale (mRS) score ≥2, recurrent stroke, changes in MoCA score, and changes in VaDAS-Cog score.

Secondary endpoints include additional functional and cognitive assessments at 24 and 52 weeks, as well as MRI markers of white matter hyperintensities, new infarctions, microbleeds, and brain atrophy. Safety assessments will include adverse events (AEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs).

The study aims to determine whether Edaravone Dexborneol Sublingual Tablets improve functional outcomes and cognitive performance in patients with small vessel disease-related stroke.

DETAILED DESCRIPTION:
This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial evaluating the efficacy and safety of Edaravone Dexborneol Sublingual Tablets in patients with acute ischemic stroke due to small vessel disease (TASTE-SVD).

1. Background and Rationale Cerebral small vessel disease (CSVD) is a major contributor to stroke, cognitive decline, and disability. Currently, there are no approved targeted therapies specifically addressing the pathophysiology of CSVD-related ischemic stroke. Edaravone Dexborneol, a novel free radical scavenger and anti-inflammatory agent, has shown neuroprotective effects in preclinical models and clinical trials for ischemic stroke. The TASTE-SL trial demonstrated that Edaravone Dexborneol improved functional outcomes at 90 days in acute ischemic stroke patients.
2. Study Design and Methods A total of 600 participants will be recruited across 50 clinical sites in China. Participants must be 30-80 years old and have an MRI-confirmed recent small subcortical infarct (RSSI).

   Eligible participants will be randomized 1:1 into:
   * Treatment group: Edaravone Dexborneol Sublingual Tablets (Edaravone 30 mg + Dexborneol 6 mg), twice daily for 24 weeks.
   * Control group: Placebo, twice daily for 24 weeks.

   Following the 24-week treatment period, participants will enter a 28-week follow-up phase, making the total study duration 52 weeks per participant.
3. Primary and Secondary Endpoints

Primary endpoint (Week 24): A hierarchical composite endpoint including:

1. All-cause mortality
2. Modified Rankin Scale (mRS) score ≥2
3. Recurrent stroke
4. Change in MoCA score from baseline
5. Change in VaDAS-Cog score from baseline

Secondary endpoints include (Week 24 & 52):

* Cognitive and functional assessments (MoCA, MMSE, IADL, HAMD, TMT-A/B)
* MRI markers of disease progression (e.g., white matter hyperintensities, infarct burden, microbleeds, brain atrophy)
* Safety outcomes, including adverse events (AEs), treatment-related AEs (TRAEs), and serious AEs (SAEs).

  4. Statistical Analysis The primary analysis will use the Win Ratio method to compare hierarchical composite endpoints between treatment groups. Secondary endpoints will be analyzed using Cochran-Mantel-Haenszel tests (for categorical outcomes) and Mixed-Effect Models for Repeated Measures (MMRM) (for continuous outcomes).

  5. Significance This study aims to determine whether Edaravone Dexborneol Sublingual Tablets can improve functional outcomes, prevent cognitive decline, and reduce stroke recurrence in CSVD-related ischemic stroke. If successful, the findings may support a new treatment approach for this high-risk population.

ELIGIBILITY:
1. Inclusion Criteria:

1. Age: Between 30 and 80 years .
2. MRI-confirmed recent small subcortical infarct (RSSI): A lesion in the small penetrating artery territory, detected as DWI hyperintensity and ADC hypointensity, with a maximum axial diameter ≤20 mm.
3. White Matter Hyperintensity (WMH) Burden: Fazekas score ≥2 (total score range: 0-6).
4. Time from Stroke Onset: ≤3 weeks from symptom onset to randomization.
5. Pre-stroke Functional Status: Modified Rankin Scale (mRS) ≤1 before the index stroke.
6. Cognitive Function: No prior diagnosis of cognitive impairment or dementia.
7. Education Level: At least primary school education and capable of completing cognitive assessments as judged by the investigator.
8. Contraception Requirements:Women of childbearing potential and male participants with female partners of childbearing potential must agree to use effective contraception during the study and 30 days after the last dose of the investigational drug.Female participants must have a negative pregnancy test before enrollment.
9. Informed Consent: Participants or their legal representatives must voluntarily sign an informed consent form (ICF).

2. Exclusion Criteria:

1. Intracranial Hemorrhagic Diseases: Evidence of hemorrhagic stroke, epidural hematoma, subarachnoid hemorrhage, or other bleeding disorders detected by head imaging (MRI/CT).However, hemorrhagic transformation may be assessed by the investigator for potential inclusion.
2. Severe Consciousness Disturbance: NIHSS item 1a score >1 (indicative of significant impairment in consciousness).
3. Cortical Infarcts or Other Brain Abnormalities:Co-existing cortical infarcts, hydrocephalus, or other non-vascular white matter diseases (e.g., multiple sclerosis, carbon monoxide poisoning-related leukoencephalopathy).
4. Severe Carotid Artery Stenosis: Requiring surgical intervention (>50% stenosis).
5. Systemic Conditions Affecting Cognition:Endocrine disorders, vitamin deficiencies, systemic autoimmune diseases that can cause cognitive impairment.
6. Neurological Disorders Associated with Cognitive Decline:CNS infections, Creutzfeldt-Jakob disease, primary Parkinson's disease, epilepsy, brain tumors, or severe traumatic brain injury.
7. Pre-existing Severe Psychiatric Disorders:Diagnosed with major depressive disorder, vascular cognitive impairment, Alzheimer's disease, Parkinson's disease dementia, Lewy body dementia, frontotemporal dementia, or any cognitive dysfunction unrelated to stroke.
8. Severe Physical Disability or Language Impairment:Severe hemiplegia or aphasia that significantly affects cognitive assessment.
9. Use of Cognitive-Enhancing Medications:Within 4 weeks prior to screening, including but not limited to:Cholinesterase inhibitors (donepezil, rivastigmine, galantamine), NMDA receptor antagonists (memantine),Other neuroprotective agents (sodium oligomannate, lecanemab)
10. Severe Liver or Kidney Dysfunction:Active liver disease (acute hepatitis, chronic active hepatitis, cirrhosis) or ALT/AST >2× ULN.
11. Severe renal impairment (serum creatinine >1.5× ULN).
12. Life Expectancy <1 year due to severe systemic diseases.
13. Contraindications to MRI:Participants with MRI-incompatible implants, severe claustrophobia, or inability to undergo MRI.
14. Known Allergies:History of hypersensitivity to Dexborneol, natural borneol, edaravone, or any excipients (e.g., mannitol, copovidone, microcrystalline cellulose, silica, magnesium stearate).
15. Pregnancy and Lactation:Pregnant or lactating women, or those planning pregnancy during the study period.
16. Participation in Other Clinical Trials:Enrolled in another clinical trial within the last 30 days.
17. Other Investigator-Determined Factors:Any other medical, psychological, or social condition that, in the investigator's judgment, makes the patient unsuitable for participation.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2027-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Hierarchical Composite Endpoint | 24 weeks
  This composite outcome consists of five hierarchical endpoints at 24 weeks, analyzed using the Win Ratio method:
  1. All-Cause Mortality
  2. Modified Rankin Scale (mRS) Score ≥2
  3. Stroke Recurrence
  4. Change in Montreal Cognitive Assessment (MoCA) Score from Baseline
  5. Change in Vascular Dementia Assessment Scale-Cognitive Subscale (VaDAS-Cog) Score from Baseline The Win Ratio approach will be used to analyze these outcomes in order of priority.
All-Cause Mortality | 24weeks
  The number of participants who experience all-cause mortality at 24 weeks. All-cause mortality includes death from any reason, such as cardiovascular, neurological, or other systemic causes. This measure is used to assess the overall survival impact of the intervention.
Modified Rankin Scale (mRS) Score ≥2 | 24 weeks
  The proportion of participants with a modified Rankin Scale (mRS) score ≥2 at 24 weeks. The mRS is a widely used functional outcome measure that assesses the degree of disability or dependence in daily activities following a stroke. The scale ranges from 0 (no symptoms) to 6 (death), with scores of 2 or higher indicating functional dependence. A higher proportion of participants with mRS ≥2 suggests a worse functional outcome.
Stroke Recurrence | 24 weeks
  The number of participants who experience a recurrent stroke within 24 weeks of treatment. Recurrent stroke is defined as a new ischemic or hemorrhagic stroke occurring after the initial qualifying event, confirmed by neurological symptoms lasting ≥24 hours and neuroimaging evidence (MRI or CT). This measure assesses the effectiveness of the intervention in preventing subsequent strokes
Change in Montreal Cognitive Assessment (MoCA) Score from Baseline | 24 weeks
  The change in Montreal Cognitive Assessment (MoCA) scores from baseline to 24 weeks of treatment. The MoCA is a cognitive screening tool that assesses multiple domains, including attention, concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive function. A greater positive change from baseline represents an improvement in cognitive function.
Change in Vascular Dementia Assessment Scale-Cognitive Subscale (VaDAS-Cog) Score from Baseline | 24 weeks
  The change in Vascular Dementia Assessment Scale-Cognitive Subscale (VaDAS-Cog) score from baseline to 24 weeks of treatment. The VaDAS-Cog is a neuropsychological assessment tool specifically designed to evaluate cognitive impairments associated with vascular dementia. VaDAS-Cog was created by adding five subtests to the ADAS-Cog that reflect attention and executive functions. The total score ranges from 0 to 70, with lower scores indicating lesser severity.

SECONDARY OUTCOMES:
All cause mortality | 24 weeks
  The number of participants who experience all-cause mortality at 24 weeks. All-cause mortality includes death from any reason, such as cardiovascular, neurological, or other systemic causes. This measure is used to assess the overall survival impact of the intervention.
Modified Rankin Scale (mRS) Score ≥2 | 24 weeks
  The proportion of participants with a modified Rankin Scale (mRS) score ≥2 at 24 weeks. The mRS is a widely used functional outcome measure that assesses the degree of disability or dependence in daily activities following a stroke. The scale ranges from 0 (no symptoms) to 6 (death), with scores of 2 or higher indicating functional dependence. A higher proportion of participants with mRS ≥2 suggests a worse functional outcome.
Stroke recurrence | 24 weeks
  The number of participants who experience a recurrent stroke within 24 weeks of treatment. Recurrent stroke is defined as a new ischemic or hemorrhagic stroke occurring after the initial qualifying event, confirmed by neurological symptoms lasting ≥24 hours and neuroimaging evidence (MRI or CT). This measure assesses the effectiveness of the intervention in preventing subsequent strokes
Post-stroke cognitive impairment | 24 weeks
  Number of participants with post-stroke cognitive impairment, defined as a MOCA score < 22
Cognitive function (MMSE) | 24 weeks
  Changes in Mini-Mental State Examination (MMSE) score from baseline. MMSE includes the assessment of 11 cognitive functions, which encompass orientation, registration of information, attention/calculation abilities, recall, naming, repetition, comprehension (both verbal and written), writing, and visuospatial construction skills. The MMSE scale ranges from 0 to 30 points, with higher scores indicating a better outcome.
Cognitive function (MoCA) | 24 weeks
  The change in Montreal Cognitive Assessment (MoCA) scores from baseline to 24 weeks of treatment. The MoCA is a cognitive screening tool that assesses multiple domains, including attention, concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive function. A greater positive change from baseline represents an improvement in cognitive function.
Cognitive function (VaDAS-Cog) | 24 weeks
  Changes in Vascular Dementia Assessment Scale-Cognitive (VaDAS-Cog) score from baseline. The VaDAS-Cog is a neuropsychological assessment tool specifically designed to evaluate cognitive impairments associated with vascular dementia. VaDAS-Cog was created by adding five subtests to the ADAS-Cog that reflect attention and executive functions. The total score ranges from 0 to 70, with lower scores indicating lesser severity.
Depression (HAMD) | 24 weeks
  Changes in Hamilton Depression Rating Scale (HAMD) score from baseline. The HAMD is a widely used clinical tool for assessing the severity of depression. It consists of multiple items that evaluate various aspects of depressive symptoms, including mood, guilt, suicidal ideation, work and interest, among others. It is scored on a scale from 0 to 52, with higher scores indicating more severe symptoms.
Activity of Daily Living | 24 weeks
  Changes in Instrumental Activities of Daily Living (IADL) score from baseline.IADL are activities that support daily life and are oriented toward interacting with your environment. Common IADLs include: Care of others; Care of pets; Child rearing; Communication management; Driving and community mobility; Financial management; Health management and maintenance; Home establishment and management; Meal preparation and clean up; Religious and spiritual activities and expressions; Safety procedure and emergency responses; Shopping. It is scored on a scale from 0 to 31, with higher scores indicating more severe symptoms.
Adverse events | 24 weeks
  Adverse events, confirmed by the Clinical Event Committee.
Serious adverse events | 24 weeks
  Serious adverse events, confirmed by the Clinical Event Committee.
Liver function impairment | 24 weeks
  Number of participants with Alanine Aminotransferase level >2.0×upper limit of the normal
Renal function impairment | 24 weeks
  Number of participants with serum creatinine >1.5×upper limit of the normal.
Composite endpoint | 24 weeks
  Composite endpoint comprising all-cause mortality, mRS ≥2, and stroke recurrence.
Change in White Matter Hyperintensity Fazekas Score from Baseline | 52 weeks
  The change in White Matter Hyperintensity (WMH) Fazekas Score from baseline to 52 weeks. The Fazekas scale is a validated measure of small vessel disease burden, ranging from 0 (no WMH) to 6 (severe WMH involvement). An increase in Fazekas score suggests disease progression, while a decrease or stabilization may indicate treatment efficacy.
Number of New MRI-Confirmed Infarcts | 52 weeks
  The number of new infarcts confirmed by MRI at 52 weeks, compared to baseline. New infarcts are defined as newly developed ischemic lesions identified on diffusion-weighted imaging (DWI) or fluid-attenuated inversion recovery (FLAIR) sequences. A higher number of new infarcts indicates increased disease progression.
Change in Number of Microbleeds from Baseline | 52 weeks
  The change in the number of microbleeds on MRI from baseline to 52 weeks, assessed using susceptibility-weighted imaging (SWI) or T2-weighted gradient-echo imaging*. Microbleeds are markers of cerebral small vessel disease and increased burden may indicate worsening vascular pathology.
Change in White Matter Hyperintensity Volume from Baseline | 52 weeks
  The change in White Matter Hyperintensity (WMH) volume from baseline to 52 weeks, assessed using quantitative MRI analysis. This measure is to evaluate the impact of treatment on the progression of small vessel disease. A decrease in WMH volume suggests treatment efficacy.
Change in Brain Atrophy Index from Baseline | 52 weeks
  The change in Brain Atrophy Index from baseline to 52 weeks, measured using MRI volumetric analysis. Brain atrophy is associated with cognitive decline and small vessel disease progression. A higher atrophy index suggests neurodegeneration, while stabilization or a slower rate of change may indicate treatment benefit
All cause mortality | 52weeks
  The number of participants who experience all-cause mortality at 24 weeks. All-cause mortality includes death from any reason, such as cardiovascular, neurological, or other systemic causes. This measure is used to assess the overall survival impact of the intervention.
Modified Rankin Scale (mRS) Score ≥2 | 52weeks
  The proportion of participants with a modified Rankin Scale (mRS) score ≥2 at 24 weeks. The mRS is a widely used functional outcome measure that assesses the degree of disability or dependence in daily activities following a stroke. The scale ranges from 0 (no symptoms) to 6 (death), with scores of 2 or higher indicating functional dependence. A higher proportion of participants with mRS ≥2 suggests a worse functional outcome.
Stroke recurrence | 52 weeks
  The number of participants who experience a recurrent stroke within 24 weeks of treatment. Recurrent stroke is defined as a new ischemic or hemorrhagic stroke occurring after the initial qualifying event, confirmed by neurological symptoms lasting ≥24 hours and neuroimaging evidence (MRI or CT). This measure assesses the effectiveness of the intervention in preventing subsequent strokes
Post-stroke cognitive impairment | 52weeks
  Number of participants with post-stroke cognitive impairment, defined as a MOCA score < 22
Cognitive function (MMSE) | 52weeks
  Changes in Mini-Mental State Examination (MMSE) score from baseline. MMSE includes the assessment of 11 cognitive functions, which encompass orientation, registration of information, attention/calculation abilities, recall, naming, repetition, comprehension (both verbal and written), writing, and visuospatial construction skills. The MMSE scale ranges from 0 to 30 points, with higher scores indicating a better outcome.
Cognitive function (MoCA) | 52weeks
  The change in Montreal Cognitive Assessment (MoCA) scores from baseline to 24 weeks of treatment. The MoCA is a cognitive screening tool that assesses multiple domains, including attention, concentration, executive function, memory, language, visuospatial skills, abstract thinking, calculation, and orientation. Scores range from 0 to 30, with higher scores indicating better cognitive function. A greater positive change from baseline represents an improvement in cognitive function.
Cognitive function (VaDAS-Cog) | 52weeks
  Changes in Vascular Dementia Assessment Scale-Cognitive (VaDAS-Cog) score from baseline. The VaDAS-Cog is a neuropsychological assessment tool specifically designed to evaluate cognitive impairments associated with vascular dementia. VaDAS-Cog was created by adding five subtests to the ADAS-Cog that reflect attention and executive functions. The total score ranges from 0 to 70, with lower scores indicating lesser severity.
Depression (HAMD) | 52weeks
  Changes in Hamilton Depression Rating Scale (HAMD) score from baseline. The HAMD is a widely used clinical tool for assessing the severity of depression. It consists of multiple items that evaluate various aspects of depressive symptoms, including mood, guilt, suicidal ideation, work and interest, among others. It is scored on a scale from 0 to 52, with higher scores indicating more severe symptoms.
Activity of Daily Living | 52weeks
  Changes in Instrumental Activities of Daily Living (IADL) score from baseline.IADL are activities that support daily life and are oriented toward interacting with your environment. Common IADLs include: Care of others; Care of pets; Child rearing; Communication management; Driving and community mobility; Financial management; Health management and maintenance; Home establishment and management; Meal preparation and clean up; Religious and spiritual activities and expressions; Safety procedure and emergency responses; Shopping. It is scored on a scale from 0 to 31, with higher scores indicating more severe symptoms
Adverse events | 52weeks
  Adverse events, confirmed by the Clinical Event Committee.
Serious adverse events | 52weeks
  Serious adverse events, confirmed by the Clinical Event Committee.
Liver function impairment | 52weeks
  Number of participants with Alanine Aminotransferase level >2.0×upper limit of the normal
Renal function impairment | 52weeks
  Number of participants with serum creatinine >1.5×upper limit of the normal.
Composite endpoint | 52weeks
  Composite endpoint comprising all-cause mortality, mRS ≥2, and stroke recurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu Y, Wang A, Tang R, Li S, Tian X, Xia X, Ren J, Yang S, Chen R, Zhu S, Feng X, Yao J, Wei Y, Dong X, Ling Y, Yi F, Deng Q, Guo C, Sui Y, Han S, Wen G, Li C, Dong A, Sun X, Wang Z, Shi X, Liu B, Fan D. Sublingual Edaravone Dexborneol for the Treatment of Acute Ischemic Stroke: The TASTE-SL Randomized Clinical Trial. JAMA Neurol. 2024 Feb 19;81(4):319-26. doi: 10.1001/jamaneurol.2023.5716. Online ahead of print. PMID 38372981
- [Background] Xu J, Wang Y, Wang A, Gao Z, Gao X, Chen H, Zhou J, Zhao X, Wang Y. Safety and efficacy of Edaravone Dexborneol versus edaravone for patients with acute ischaemic stroke: a phase II, multicentre, randomised, double-blind, multiple-dose, active-controlled clinical trial. Stroke Vasc Neurol. 2019 Apr 22;4(3):109-114. doi: 10.1136/svn-2018-000221. eCollection 2019 Sep. PMID 31709115
- [Background] Xu J, Wang A, Meng X, Yalkun G, Xu A, Gao Z, Chen H, Ji Y, Xu J, Geng D, Zhu R, Liu B, Dong A, Mu H, Lu Z, Li S, Zheng H, Chen X, Wang Y, Zhao X, Wang Y; TASTE Trial Investigatorsdagger. Edaravone Dexborneol Versus Edaravone Alone for the Treatment of Acute Ischemic Stroke: A Phase III, Randomized, Double-Blind, Comparative Trial. Stroke. 2021 Mar;52(3):772-780. doi: 10.1161/STROKEAHA.120.031197. Epub 2021 Feb 16. PMID 33588596